CLINICAL TRIAL: NCT00701935
Title: Effect of Exenatide on Abdominal Fat Distribution in Patients With Type 2 Diabetes Pretreated With Metformin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment was much slower than anticipated, leading to a decision to terminate the study early for enrollment futility.
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-CA-GWCE
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2013-02-13 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental)
  Interventions: Drug: exenatide

INTERVENTIONS:
Drug: placebo — subcutaneous injection, twice a day
  Arms: 1
Drug: exenatide — subcutaneous injection, twice a day, 10mcg
  Arms: 2

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled trial will assess the effects of twice-daily subcutaneous injection with exenatide versus treatment with matching placebo injection on abdominal visceral fat content.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 85 years of age, inclusive.
* Patients with type 2 diabetes
* Patients have been treated with metformin, at a stable dose for at least 3 months prior to Visit 1
* Patients have HbA1c of 7.0% to 8.9%, inclusive.
* Patients have a body mass index >27 kg/m2 and <40 kg/m2 and meet local CT scan body weight requirements. For South Asian, Japanese, and Chinese patients, a body mass index >=25 kg/m2 is acceptable as the lower limit.
* Patients have a history of stable body weight (not varying by >2 kg in the 3 months prior to Visit 1).
* Medications for the treatment of high blood pressure are stable with respect to treatment regimen for 4 weeks prior to Visit 1.
* Stable regimen of lipid-lowering agents for 6 weeks prior to Visit 1.

Exclusion Criteria:

* Have received treatment in the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have an active or untreated malignancy, or have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years.
* Have a history of renal transplantation, or are currently receiving renal dialysis.
* Have had a clinically significant history of cardiac disease or presence of active cardiac disease within 1 year prior to Visit 1, including myocardial infarction, clinically significant arrhythmia, unstable angina, moderate to severe congestive heart failure, coronary artery bypass surgery, or angioplasty; or is expected to require coronary artery bypass surgery or angioplasty during the course of the study.
* Have known hemoglobinopathy or clinically significant, chronic anemia.
* Known or are likely to become transfusion dependent during the study.
* Have active, symptomatic proliferative retinopathy.
* Are receiving chronic treatment for gastrointestinal disease with a drug directly affecting gastrointestinal motility. (i.e. metoclopramide, cisapride, and chronic use of macrolide antibiotics)
* Have severe gastrointestinal disease, including gastroparesis.
* Are receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within 2 months immediately prior to Visit 1.
* Have taken exenatide, liraglutide or any other GLP-1 receptor agonist in the past 6 months, either in a clinical study or as commercially available medication. Patients with known allergy to exenatide should be excluded.
* Have used any prescription or over the counter drug to promote weight loss within 3 months prior to Visit 1, or intend to use such a drug during the study. (Examples: Xenical [orlistat], Meridia [sibutramine], Acutrim [phenylpropanolamine], Acomplia [rimonabant]).
* Have participated in a structured weight loss program within 3 months prior to Visit 1, or intend to participate in such a plan during this study.
* Have been treated for longer than 2 weeks with any of the following excluded medications within 3 months prior to Visit 1: Insulin; Thiazolidinediones; Alpha-glucosidase inhibitors; Sulfonylureas; Oral DPP-IV inhibitors; Meglitinides.
* Are taking warfarin, or a coumarol derivative.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD Eli Lilly and Company, Study Director — Eli Lilly and Company
Locations (17):
- United States (5):
  - Research Site, Temple, Arizona
  - Research Site, Colorado Springs, Colorado
  - Research Site, Honolulu, Hawaii
  - Research Site, Bellevue, Nebraska
  - Research Site, Las Vegas, Nevada
- Canada (12):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Saint John, New Brunswick
  - Research Site, Brampton, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial planned enrolment was 12 months, starting August 2008. Eventual enrolment time was 3+ years - decision made to close end of 2011.
  Number of patients initially planned: 94 randomized and 74 completers Final number of patients: 80 randomized and 53 completers
Groups:
- Exenatide BID: Subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for remainder of 6 months)
- Placebo: Subcutaneous injection of placebo twice a day for 6 months
Period: Overall Study
Arm/Group | Exenatide BID | Placebo
Started | 43 | 37
Completed | 27 | 26
Not Completed | 16 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide BID | Placebo | Total
Number analyzed (Participants) | 43 | 37 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (12.2) | 57.9 (11.0) | 58.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 23 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Abdominal Visceral Fat From Baseline to 6 Months
Description: Percentage change in abdominal visceral fat
Time Frame: baseline, 6 months
Population: Primary analysis done on the Intent To Treat (ITT) Population including all randomized patients receiving at least one dose of study drug according to the treatment the subjects are randomized to regardless of what study drug patients received
Measure: Least Squares Mean (Standard Error); unit: % change
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 29 | 27
% change | -5.28 (3.23) | -4.30 (3.53)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; The power calculation is based on a two-sided t-test and significance level of 0.05. Hypotheses for sample size: Power: 80% Drop-out rate: 20% Difference in the percentage change in abdominal visceral fat from baseline to 6 months between exenatide and placebo: 10% Common standard deviation: 15% 94 patients are needed to attain the 37 patients randomized and analyzed in each group; Test type: Superiority or Other; p = 0.8252, ANCOVA — p-values were not adjusted for multiple comparisons; The ANCOVA model includes terms of treatment, gender, investigator and baseline abdominal visceral fat; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-9.92 to 7.95], Standard Error of Mean 4.432

2. Secondary Outcome: Percentage Change in Total Abdominal Fat From Baseline to 6 Months
Description: Percentage change in total abdominal fat
Time Frame: baseline, 6 months
Population: Analysis done on the ITT Population including all randomized patients receiving at least one dose of study drug according to the treatment the subjects are randomized to regardless of what study drug patients received
Measure: Least Squares Mean (Standard Error); unit: % change
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 26 | 25
% change | -5.81 (2.28) | -3.74 (2.36)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Superiority or Other; p = 0.5207, ANCOVA — p-values were not adjusted for multiple comparisons; The ANCOVA model includes terms of treatment, gender, investigator and baseline total abdominal fat; Mean Difference (Final Values) = -2.07, 95% CI 2-sided [-8.53 to 4.39], Standard Error of Mean 3.193

3. Secondary Outcome: Percentage Change in Subcutaneous Abdominal Fat From Baseline to 6 Months
Description: Percentage change in subcutaneous abdominal fat
Time Frame: baseline, 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: % change
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 25 | 25
% change | -7.27 (1.93) | -3.56 (1.97)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Superiority or Other; p = 0.1755, ANCOVA — p-values were not adjusted for multiple comparisons; The ANCOVA model includes terms of treatment, gender, investigator and baseline subcutaneous abdominal fat; Mean Difference (Final Values) = -3.71, 95% CI 2-sided [-9.15 to 1.73], Standard Error of Mean 2.687

4. Secondary Outcome: Change in HbA1c From Baseline to 6 Months
Description: Change in HbA1c from baseline to 6 months. HbA1c is a measurement of the amount of hemogobin that is glycosylated.
Time Frame: baseline, 6 months
Population: Analysis done on the ITT Population including all randomized patients receiving at least one dose of study drug according to the treatment the subjects are randomized to regardless of what study drug patients received. Last observation (month 6 or early discontinuation) was analysed.
Measure: Least Squares Mean (Standard Error); unit: % change
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 42 | 33
% change | -0.69 (0.12) | 0.19 (0.15)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-values were not adjusted for multiple comparisons; ANCOVA analysis included the following factors: treatment, gender, investigator and baseline HbA1c; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-1.19 to -0.57], Standard Error of Mean 0.155

5. Secondary Outcome: Percentage of Patients With HbA1c <=7.0% at 6 Months
Description: Percentage of patients with HbA1c values <= 7.0% measured at 6 months. HbA1c is a measurement of the amount of hemogobin that is glycosylated.
Time Frame: 6 months
Population: Analysis done on the ITT Population including all randomized patients receiving at least one dose of study drug according to the treatment the subjects are randomized to regardless of what study drug patients received.Analysis done only for patients with measurement at Month 6.
Measure: Number; unit: Percentage of patients
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 28 | 28
Percentage of patients | 60.7 | 21.4

6. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to 6 Months
Description: Change in Fasting plasma glucose
Time Frame: baseline, 6 months
Population: Analysis done on the ITT Population including all randomized patients receiving at least one dose of study drug according to the treatment the subjects are randomized to regardless of what study drug patients received. Analysis done only for patients with measurement at Month 6.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 26 | 26
mmol/L | -1.47 (0.36) | -0.08 (0.38)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Superiority or Other; p = 0.0073, ANCOVA — p-values were not adjusted for multiple comparisons; The ANCOVA model includes terms of treatment, gender, investigator and baseline fasting plasma glucose; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-2.38 to -0.40], Standard Error of Mean 0.491

7. Secondary Outcome: Change in Weight From Baseline to 6 Months
Description: Change in weight
Time Frame: baseline, 6 months
Population: Analysis done on the ITT Population including all randomized patients receiving at least one dose of study drug according to the treatment the subjects are randomized to regardless of what study drug patients received. Last observation (month 6 or early discontinuation) was analyzed.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 42 | 33
kg | -2.54 (0.57) | -0.33 (0.72)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Superiority or Other; p = 0.0035, ANCOVA — p-values were not adjusted for multiple comparisons; The ANCOVA model includes terms of treatment, gender, investigator and baseline body weight; Mean Difference (Final Values) = -2.21, 95% CI 2-sided [-3.66 to -0.76], Standard Error of Mean 0.725

8. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to 6 Months
Description: Change in Systolic blood pressure
Time Frame: baseline, 6 months
Population: Analysis done on the ITT Population including all randomized patients receiving at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 29 | 28
mmHg | -7.48 (12.57) | 1.79 (12.41)

9. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to 6 Months
Description: Change in Diastolic blood pressure
Time Frame: baseline, 6 months
Population: Analysis done on the ITT Population including all randomized patients receiving at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 29 | 28
mmHg | -2.86 (6.99) | -0.18 (8.97)

10. Secondary Outcome: Change in Total Cholesterol From Baseline to 6 Months
Description: Change in total cholesterol
Time Frame: baseline, 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 29 | 27
mmol/L | -0.06 (0.18) | 0.14 (0.20)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Superiority or Other; p = 0.4145, ANCOVA — p-values were not adjusted for multiple comparisons; The ANCOVA model includes terms of treatment, gender, investigator and baseline total cholesterol; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.71 to 0.30], Standard Error of Mean 0.248

11. Secondary Outcome: Change in Triglycerides From Baseline to 6 Months
Description: Change in triglycerides
Time Frame: baseline, 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 29 | 27
mmol/L | -0.17 (0.21) | 0.06 (0.23)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Superiority or Other; p = 0.4007, ANCOVA — p-values were not adjusted for multiple comparisons; The ANCOVA model includes terms of treatment, gender, investigator and baseline triglycerides; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.80 to 0.33], Standard Error of Mean 0.279

12. Secondary Outcome: Change in High-Density Lipoprotein (HDL) Cholesterol From Baseline to 6 Months
Description: Change in HDL cholesterol
Time Frame: baseline, 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 29 | 27
mmol/L | 0.06 (0.04) | 0.04 (0.04)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Superiority or Other; p = 0.7915, ANCOVA — p-values were not adjusted for multiple comparisons; The ANCOVA model includes terms of treatment, gender, investigator and baseline HDL cholesterol; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.08 to 0.11], Standard Error of Mean 0.048

13. Secondary Outcome: Assessment of Event Rate of Treatment- Emergent Hypoglycemic Event
Description: All hypoglycemia episodes defined as major (results in loss of consciousness, seizure or coma resolving after administration of glucagon or glucose OR needing third-party assistance to resolve due to severe impairment in consciousness and associated with glucose concentration < 2.8 mol/L.) or minor (non-major event with symptoms consistent with hypoglycemia and glucose value < 2.8 mmol/L prior to treating) or symptoms of hypoglycemia (does not meet the criteria for a major or minor event).
Time Frame: baseline, 6 months
Population: Analysis done on the ITT Population including all randomized patients receiving at least one dose of study drug.
Measure: Mean (Standard Error); unit: hypoglycemia rate/year
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 43 | 37
hypoglycemia rate/year | 0.41 (0.15) | 0.12 (0.09)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Event rate per subject year was calculated for each subject : (number of events observed from a subject/exposure from a subject)*365.25 where exposure = last post-baseline visit date - baseline visit date; Test type: Superiority or Other; p = 0.1388, Regression, Linear — p-values were not adjusted for multiple comparisons; Generalized linear model was used with the assumption of an underlying Poisson distribution and the logarithm of exposure (years) as offset variable; Ratio = 3.28, 95% CI 2-sided [0.68 to 15.77], Standard Error of Mean 2.63

ADVERSE EVENTS:
Arm/Group | Exenatide BID | Placebo
Serious Adverse Events (participants affected / at risk) | 3/43 | 1/37
Other Adverse Events (participants affected / at risk) | 38/43 | 25/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide BID (N=43) | Placebo (N=37)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mesenteritis (Gastrointestinal disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide BID (N=43) | Placebo (N=37)
vertigo (Ear and labyrinth disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 15 | 11
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Vomiting (Gastrointestinal disorders) | 7 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 6
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 5 | 1
Injection site reaction (General disorders) | 2 | 2
Nasopharyngitis (Infections and infestations) | 8 | 7
Influenza (Infections and infestations) | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 8 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Headache (Nervous system disorders) | 6 | 5
Dizziness (Nervous system disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
The dropout rate in the study was higher than anticipated (of 80 patients randomized, only 53 completed Study Period II), and enrollment was much slower than anticipated, leading to a decision to terminate the study early for enrollment futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No